CLINICAL TRIAL: NCT00396227
Title: A Multi-center, Randomized, Open-label, Active Controlled, Parallel Arm Study to Compare the Efficacy of 12 Weeks of Treatment With Vildagliptin 100 mg, qd to Thiazolidinedione (TZD) as add-on Therapy in Patients With Type 2 Diabetes Inadequately Controlled With Metformin Monotherapy in a Community-based Practice Setting.
Brief Title: Safety and Efficacy of Vildagliptin vs. Thiazolidinedione as add-on Therapy to Metformin in Patients With Type 2 Diabetes Not Controlled With Metformin Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLAF237A23119
Record Dates: First submitted 2006-11-02; First posted 2006-11-06 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; vildagliptin; hemoglobin A1c; metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; 2,4-thiazolidinedione; Pioglitazone; Rosiglitazone

ARMS (2):
- 1 (Experimental): Vildagliptin 100mg + Met
  Interventions: Drug: vildagliptin
- TZD (Active Comparator): TZD + metformin
  Interventions: Drug: thiazolidinedione (TZD)

INTERVENTIONS:
Drug: vildagliptin — vildagliptin as add-on to metformin
  Other Names: Galvus
  Arms: 1
Drug: thiazolidinedione (TZD) — TZD add-on to metformin
  Other Names: Actos (pioglitazone), Avandia (rosiglitazone)
  Arms: TZD

SUMMARY:
This study is designed to evaluate, in a primary care setting, the safety and efficacy of vildaglipgtin as add on therapy to metformin relative to TZD added to metformin in patients with type 2 diabetes inadequately controlled by metformin alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have received a stable dose of metformin consisting of at least 1,000 mg/day for four weeks prior to Visit 1 (week-2)
* Agreement to maintain the same dose of metformin from screening to the end of the study
* Age in the range of 18-80 years
* Body mass index (BMI) in the range of 22-40 kg/m2
* HbA1c in the range of 7.0 to 10%
* FPG <270 mg/dL (15 mmol/L)

Exclusion Criteria:

* A history of type 1 diabetes
* Liver disease
* Treatment with insulin or any oral anti-diabetic other than metformin, within 8 weeks prior to Visit 1

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 2665 (Actual)
Dates: Start 2006-10; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HemoglobinA1c (HbA1c) | after 12 weeks of treatment

SECONDARY OUTCOMES:
Change from baseline in body weight | after 12 weeks of treatment
Change from baseline in fasting plasma glucose (FPG) | after 12 weeks of treatment
Incidence of prespecified adverse events while on treatment with study drug | 12 week treatment duration

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States

REFERENCES:
- [Result] Blonde L, Dagogo-Jack S, Banerji MA, Pratley RE, Marcellari A, Braceras R, Purkayastha D, Baron M. Comparison of vildagliptin and thiazolidinedione as add-on therapy in patients inadequately controlled with metformin: results of the GALIANT trial--a primary care, type 2 diabetes study. Diabetes Obes Metab. 2009 Oct;11(10):978-86. doi: 10.1111/j.1463-1326.2009.01080.x. Epub 2009 Jul 13. PMID 19614942